CLINICAL TRIAL: NCT00731783
Title: Household vs. Individual Approach to Decolonization of Community-acquired Methicillin-resistant Staphylococcus Aureus.
Brief Title: Staphylococcus Aureus Decolonization Study
Acronym: SuDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Stephanie A. Fritz, Assistant Professor of Pediatrics, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3177 38145
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Staphylococcal Skin Infections; Abscesses; Furunculosis; Staphylococcus Aureus; MRSA Infection
Keywords: Abscesses; Furunculosis; Staphylococcus aureus colonization; Staphylococcal Skin Infections; MRSA
MeSH Terms: conditions — Staphylococcal Skin Infections; Abscess; Furunculosis; Staphylococcal Infections | interventions — Mupirocin; chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Index patient only (Active Comparator): Only the child recently treated for a skin or soft tissue infection will undergo the decolonization regimen.
  Interventions: Drug: 2% Mupirocin Ointment; Drug: 4% Chlorhexidine liquid soap; Behavioral: Hygiene protocol
- Household (Active Comparator): All members of the household (over the age of 6 months) will be asked to follow the study protocol.
  Interventions: Drug: 2% Mupirocin Ointment; Drug: 4% Chlorhexidine liquid soap; Behavioral: Hygiene protocol

INTERVENTIONS:
Drug: 2% Mupirocin Ointment — Apply ointment to the anterior nares twice daily for 5 days.
  Other Names: Bactroban
Drug: 4% Chlorhexidine liquid soap — Bathe with liquid soap daily for 5 days.
  Other Names: Hibiclens
Behavioral: Hygiene protocol — Follow key hygiene tips indefinitely. Tips are:
  * Throw out all lotions or creams that you dip your hands into and replace with pumps or pour bottles.
  * Use liquid(pour or pump) soaps instead of bar soaps.
  * Wash hands frequently or use hand sanitizer(with more than %60 alcohol) such as Germ-X or Purell.
  * Do not share personal care items such as razors and brushes.
  * Wash all sheets and towels in hot water. Wash sheets every week.
  * Use towels and wash cloths only once before washing and do not share.

SUMMARY:
The purpose of this study is to determine whether measures to eliminate the Staph germ from the skin of the index patient (with a special ointment and soap) are more effective when performed by everyone in the household rather than the patient alone, and whether these methods are effective in preventing future Staph infections. The investigators hypothesize that there will be a greater number of households who are successful in eradicating the staph germ from the index patient when all members of the household participate than households where only the index patient is treated.

DETAILED DESCRIPTION:
Methicillin-resistant Staphylococcus aureus (MRSA) was once uniformly associated with hospital-acquired infections; however, MRSA strains have emerged that thrive outside the hospital environment, causing significant morbidity and mortality among immunocompetent individuals, leading to their designation as community-acquired methicillin resistant Staphylococcus aureus (CA-MRSA).

CA-MRSA has become a major source of morbidity and mortality in our pediatric population. An important prerequisite for S. aureus infection may be nasal carriage of the organism. A variety of decolonization strategies have been used for infection prophylaxis, primarily in patients undergoing hemodialysis or surgery, with varying results. However, there are no published randomized eradication trials evaluating the decolonization and prevention of CA-MRSA infections in immunocompetent children in the outpatient setting. While the transmission of CA-MRSA within households has been reported, its contribution to recurrent CA-MRSA infection among household members is undetermined. The investigators hypothesize that spread of CA-MRSA among household members leads to recolonization or failure of decolonization in children undergoing eradication efforts.

Specific Aim: In pediatric patients presenting with a MRSA skin or soft tissue infection, compare the effectiveness of decolonization measures performed by an entire household in comparison to measures directed at the index patient alone. The investigators will conduct a randomized, controlled trial to test the hypothesis that decolonization measures performed by the entire household, specifically application of intranasal mupirocin ointment and bathing with chlorhexidine liquid soap, in addition to education and basic hygiene interventions, will be twice as effective in eradicating CA-MRSA carriage in the index patient than if the measures are performed only by the index patient.

ELIGIBILITY:
Inclusion Criteria:

Screening:

* Children aged 6 months to 21 years presenting with an active skin or soft tissue infection.

Enrollment:

* Positive MRSA culture from the abscess and from either the axilla, anterior nares or groin area (signifying both infection and colonization with MRSA).

Exclusion Criteria:

* Infants less than 6 months of age
* Dialysis or residence in a long term care facility over the past year
* Use of chlorhexidine or mupirocin in the past one month
* Pregnancy
* Immunodeficiency
* History of an adverse reaction to chlorhexidine or mupirocin.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 183 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Fritz, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Fritz SA, Hogan PG, Hayek G, Eisenstein KA, Rodriguez M, Epplin EK, Garbutt J, Fraser VJ. Household versus individual approaches to eradication of community-associated Staphylococcus aureus in children: a randomized trial. Clin Infect Dis. 2012 Mar;54(6):743-51. doi: 10.1093/cid/cir919. Epub 2011 Dec 23. PMID 22198793

RESULTS

PARTICIPANT FLOW:
Groups:
- Index Patient Only: Only the child recently treated for a skin or soft tissue infection will undergo the decolonization regimen, which includes application of 2% Mupirocin Ointment to the anterior nares twice daily for 5 days and washing with 4% Chlorhexidine liquid soap daily for 5 days.
- Household: All members of the household (over the age of 6 months) will be asked to follow the study protocol, which includes application of 2% Mupirocin Ointment to the anterior nares twice daily for 5 days and washing with 4% Chlorhexidine liquid soap daily for 5 days.
Period: One Month Follow-Up Visit
Arm/Group | Index Patient Only | Household
Started | 92 | 91
Completed | 78 | 69
Not Completed | 14 | 22
Not completed — Lost to Follow-up | 14 | 22
Period: Three Month Follow-Up Visit
Arm/Group | Index Patient Only | Household
Started | 79 | 73
Completed | 72 | 57
Not Completed | 7 | 16
Not completed — Lost to Follow-up | 7 | 16
Period: Six Month Follow-Up Visit
Arm/Group | Index Patient Only | Household
Started | 77 | 67
Completed | 71 | 64
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 6 | 3
Period: 12 Month Follow-Up Visit
Arm/Group | Index Patient Only | Household
Started | 74 | 65
Completed | 68 | 58
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Index Patient Only | Household | Total
Number analyzed (Participants) | 92 | 91 | 183
Age Continuous [Mean (Standard Deviation); unit: Years] | 6.3 (5.7) | 5.7 (6.0) | 6.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 51 | 106
  Male | 37 | 40 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Index Patients Eradicated of S. Aureus Carriage - 1 Month After Performing Decolonization Measures
Description: Eradication is defined as the absence of S. aureus carriage at the 3 sampled body sites (anterior nares, axilla, inguinal folds) of the index patient.
Time Frame: 1 month after enrollment.
Population: Modified intention to treat analysis
Measure: Number; unit: Participants
Arm/Group | Index Patient Only | Household
Number analyzed (Participants) | 78 | 69
Participants | 39 | 35
Statistical Analysis 1: Comparison: Index Patient Only vs Household; Test type: Superiority or Other; p = 1.00, Fisher Exact; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.54 to 1.97]

2. Secondary Outcome: Number of Index Patients Eradicated of S. Aureus Carriage - 3 Month After Performing Decolonization Measures
Description: as for outcome 1
Time Frame: 3 month after enrollment.
Population: Modified intention to treat analysis
Measure: Number; unit: Participants
Arm/Group | Index Patient Only | Household
Number analyzed (Participants) | 72 | 57
Participants | 39 | 41
Statistical Analysis 1: Comparison: Index Patient Only vs Household; Test type: Superiority or Other; p = 0.05, Fisher Exact; Odds Ratio (OR) = 2.17, 95% CI 2-sided [1.03 to 4.55]

3. Secondary Outcome: Number of Index Patients Eradicated of S. Aureus Carriage - 6 Month After Performing Decolonization Measures
Description: as for outcome 1
Time Frame: 6 month after enrollment.
Population: Modified intention to treat analysis
Measure: Number; unit: Participants
Arm/Group | Index Patient Only | Household
Number analyzed (Participants) | 71 | 64
Participants | 39 | 31
Statistical Analysis 1: Comparison: Index Patient Only vs Household; Test type: Superiority or Other; p = 0.49, Fisher Exact; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.39 to 1.52]

4. Secondary Outcome: Number of Index Patients Eradicated of S. Aureus Carriage - 12 Month After Performing Decolonization Measures
Description: as for outcome 1
Time Frame: 12 month after enrollment.
Population: Modified intention to treat analysis
Measure: Number; unit: Participants
Arm/Group | Index Patient Only | Household
Number analyzed (Participants) | 68 | 58
Participants | 37 | 38
Statistical Analysis 1: Comparison: Index Patient Only vs Household; Test type: Superiority or Other; p = 0.28, Fisher Exact; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.77 to 3.28]

5. Secondary Outcome: Recurrence of CA-MRSA Skin or Soft Tissue Infection - 1 Month After Enrollment.
Description: Recurrence of CA-MRSA Skin or Soft Tissue Infection
Time Frame: 1 month after enrollment
Population: Modified intention to treat analysis
Measure: Number; unit: Participants
Arm/Group | Index Patient Only | Household
Number analyzed (Participants) | 81 | 72
Participants | 21 | 11
Statistical Analysis 1: Comparison: Index Patient Only vs Household; Test type: Superiority or Other; p = 0.12, Fisher Exact; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.23 to 1.16]

6. Secondary Outcome: Recurrence of CA-MRSA Skin or Soft Tissue Infection - 3 Month After Enrollment.
Description: Recurrence of CA-MRSA Skin or Soft Tissue Infection
Time Frame: 3 month after enrollment
Population: Modified intention to treat analysis
Measure: Number; unit: Participants
Arm/Group | Index Patient Only | Household
Number analyzed (Participants) | 76 | 69
Participants | 36 | 19
Statistical Analysis 1: Comparison: Index Patient Only vs Household; Test type: Superiority or Other; p = 0.02, Fisher Exact; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.21 to 0.85]

7. Secondary Outcome: Recurrence of CA-MRSA Skin or Soft Tissue Infection - 6 Month After Enrollment.
Description: Recurrence of CA-MRSA Skin or Soft Tissue Infection
Time Frame: 6 month after enrollment
Population: Modified intention to treat analysis
Measure: Number; unit: Participants
Arm/Group | Index Patient Only | Household
Number analyzed (Participants) | 76 | 69
Participants | 46 | 26
Statistical Analysis 1: Comparison: Index Patient Only vs Household; Test type: Superiority or Other; p = 0.008, Fisher Exact; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.20 to 0.77]

8. Secondary Outcome: Recurrence of CA-MRSA Skin or Soft Tissue Infection - 12 Month After Enrollment.
Description: Recurrence of CA-MRSA Skin or Soft Tissue Infection
Time Frame: 12 month after enrollment
Population: Modified intention to treat analysis
Measure: Number; unit: Participants
Arm/Group | Index Patient Only | Household
Number analyzed (Participants) | 78 | 65
Participants | 56 | 34
Statistical Analysis 1: Comparison: Index Patient Only vs Household; Test type: Superiority or Other; p = 0.02, Fisher Exact; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.22 to 0.86]

ADVERSE EVENTS:
Time Frame: Adverse events were collected by phone approximately 7-10 days following study enrollment. The intervention only lasted 5 days and thus all adverse events would have happened by this time.
Description: There are more participants with data on adverse events than data on the primary outcome measure because some participants completed the follow-up phone call at 7-10 days (where adverse events were assessed) but failed to complete the 1 month follow-up visit (where primary outcome measure was assessed).
Arm/Group | Index Patient Only | Household
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/77
Other Adverse Events (participants affected / at risk) | 15/85 | 17/77
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Index Patient Only (N=85) | Household (N=77)
Dry Skin (Skin and subcutaneous tissue disorders) | 10 | 13
Rash (Skin and subcutaneous tissue disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No